CLINICAL TRIAL: NCT01461629
Title: Cognitive Impairment and Self-management in Adults With Heart Failure
Brief Title: Self-management and Cognitive Function in Adults With Heart Failure
Acronym: Heart ABC
Status: Completed | Type: Observational
Sponsor: Kent State University (Other)
Collaborators: Summa Health System (Other); Case Western Reserve University (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Tony Vehovec, Associate Professor, Kent State University
Other Study IDs: 10217650; 10217650 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Cognitive Impairment; Cardiac Disease; Heart Failure
Keywords: cognitive impairment; cognitive function; hospitalization; self-management; cardiac disease; heart failure
MeSH Terms: conditions — Cognitive Dysfunction; Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary sodium

GROUPS / COHORTS (1):
- heart failure: left systolic heart failure (EF </= 40%)

SUMMARY:
The purpose of this study is to assess the relationship between cognitive impairment, patient self-management, health, and health service use in adults with heart failure (NYHA Class 2 and 3). The research questions are:

1. How is cognitive impairment (memory, attention, global and executive function) related to various aspects of impaired self-management (knowledge of adherence, adherence to sodium restriction and medications, symptom monitoring of weight changes, and decision and action to seek care)?
2. How are these relationships altered when adjusting for medical, demographic, and psychosocial factors?
3. What are the relationships among degree of cognitive impairment, quality self-management, health status, and health service use?

ELIGIBILITY:
Inclusion Criteria:

* documented systolic heart failure
* NYHA class II, III of at least 6 months duration
* 50-85 years of age
* has a telephone (land line) or be willing to allow a telephone installed for duration of study

Exclusion Criteria:

* history of neurological disorder or injury
* moderate or severe head injury
* past or current history of severe psychiatric illness; specifically, psychotic disorders and bipolar disorder
* 5 year past or current history of alcohol or drug abuse
* history of learning disorder or developmental disability
* renal failure requiring dialysis
* history of sleep apnea
* current home telemonitoring program to assist w/ HF self-management
* cardiac surgery < 3 months

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50-85 years of age, documented diagnosis of systolic heart failure (EF </= 35%) at least 12 months prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2010-06; Primary Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Summa Health System, Akron, Ohio, United States

REFERENCES:
- [Derived] Kuhn TA, Gathright EC, Dolansky MA, Gunstad J, Josephson R, Hughes JW. Health Literacy, Cognitive Function, and Mortality in Patients With Heart Failure. J Cardiovasc Nurs. 2022 Jan-Feb 01;37(1):50-55. doi: 10.1097/JCN.0000000000000855. PMID 34581712
- [Derived] Walter FA, Ede D, Hawkins MAW, Dolansky MA, Gunstad J, Josephson R, Moore SM, Hughes JW. Sleep quality and daytime sleepiness are not associated with cognition in heart failure. J Psychosom Res. 2018 Oct;113:100-106. doi: 10.1016/j.jpsychores.2018.08.003. Epub 2018 Aug 10. PMID 30190041
- [Derived] Dolansky MA, Hawkins MA, Schaefer JT, Sattar A, Gunstad J, Redle JD, Josephson R, Moore SM, Hughes JW. Association Between Poorer Cognitive Function and Reduced Objectively Monitored Medication Adherence in Patients With Heart Failure. Circ Heart Fail. 2016 Dec;9(12):e002475. doi: 10.1161/CIRCHEARTFAILURE.116.002475. PMID 27895069
- [Derived] Basuray A, Dolansky M, Josephson R, Sattar A, Grady EM, Vehovec A, Gunstad J, Redle J, Fang J, Hughes JW. Dietary sodium adherence is poor in chronic heart failure patients. J Card Fail. 2015 Apr;21(4):323-9. doi: 10.1016/j.cardfail.2014.12.016. Epub 2015 Jan 7. PMID 25576680